CLINICAL TRIAL: NCT04981665
Title: Official Title ICMJE A Phase 2, Open-Label, Multi-Center, Single Arm Study to Evaluate the Efficacy and Safety of TACE Sequential Tislelizumab as Adjuvant Therapy in Participants With Hepatocellular Carcinoma Who Are at High Risk of Recurrence After Curative Hepatic Resection
Brief Title: A Study to Evaluate TACE Sequential Tislelizumab as Adjuvant Therapy in Participants With HCC at High Risk of Recurrence After Curative Resection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: First Hospital of China Medical University (Other); Shandong Cancer Hospital and Institute (Other); The Affiliated Hospital Of Southwest Medical University (Other); Hainan People's Hospital (Other); Tianjin Third Central Hospital (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-2008
Record Dates: First submitted 2021-07-25; First posted 2021-07-29 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Hepatocellular Carcinoma; Adjuvant Therapy
Keywords: Hepatocellular carcinoma; Immunotherapy; Transarterial chemoembolization; Recurrence; Antineoplastic Agents, Immunological; Antineoplastic Agents
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — tislelizumab; Immunotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postoperative TACE + Tislelizumab 200mg IV Q3W (Experimental): TACE will be performed after curative resection (4±1w) once and then Tislelizumab Injection will be initiated after TACE (5±2d). Tislelizumab will be administered every three weeks, until the disease recurrence, intolerable toxicity, death, withdrawal of consent or completion of 17 cycles of Tislelizumab.
  Interventions: Drug: Tislelizumab; Drug: TACE

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200mg IV Q3W
  Other Names: BGB-A317; Immunotherapy; Anti-PD-1 therapy
Drug: TACE — TACE will be performed after curative resection (4±1w)
  Other Names: Transarterial Chemoembolization

SUMMARY:
This is an open label, multi-center, phaseⅡstudy to evaluate the efficacy and safety of TACE sequential tislelizumab as adjuvant therapy in hepatocellular carcinoma (HCC) patients who are at high risk of recurrence after curative resection.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a malignant tumor with high morbidity and mortality. Surgical resection is the most important radical treatment. However, the recurrence rate is high especially in the patients with high risk of recurrence after curative resection. How to reduce postoperative recurrence and improve survival is currently a direction that is worth exploring.

Until now there is no standard postoperative adjuvant therapy. Previous studies have shown that TACE combined with PD-1 inhibitors has a synergistic enhancement effect, and this study is to explore the efficacy and safety of TACE sequential tislelizumab as adjuvant therapy in HCC patients who are at high risk of recurrence after curative resection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a histopathological or cytologically diagnosis of HCC
* Subjects who have undergone a curative resection
* High risk for HCC recurrence as protocol defined
* No previous systematic treatment and locoregional therapy for HCC
* Child-Pugh Score, Class A
* ECOG performance status 0 or 1
* Full recovery from surgical resection
* Adequate organ function
* Absence of major macrovascular invasion
* No extrahepatic spread
* Life expectancy of at least 6 months

Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC or mixed cholangiocarcinoma and HCC
* Evidence of residual, recurrent, or metastatic disease
* Known history of serious allergy to any monoclonal antibody
* History of hepatic encephalopathy
* Tumor thrombus in portal vein or superior mesenteric vein or inferior caval vein
* Portal hypertension with bleeding esophageal or gastric varices within 6 months prior to initiation of treatment
* Any bleeding or thrombotic disorder within 6 months prior to initiation of treatment
* Any active malignancy within 2 years prior to the start of treatment
* Active or history of autoimmune disease
* Other acute or chronic conditions, psychiatric disorders, or laboratory abnormalities that may increase the risk of study participation
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or other immunotherapy
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
2-year Recurrence Free Survival Rate (2-year RFS rate) | Observation period 24 months
  2-year RFS rate is defined as the proportion of patients alive and free of recurrence at 2 years after curative resection.

SECONDARY OUTCOMES:
Recurrence-Free Survival (RFS) | 24 months
  RFS is defined as the time from the date of curative resection to the first documented recurrence or death due to any cause, whichever occurs first.
Time to recurrence (TTR) | 24 months
  TTR is defined as the time from the date of curative resection to the first documented recurrence.
Overall Survival (OS） | 24 months
  OS is defined as the time from the date of curative resection until death due to any cause.
1-year RFS rate | 12 months
  1-year RFS rate is defined as the proportion of patients alive and free of recurrence at 1 years after curative resection.
1-year OS rate/2-year OS rate | 12 months/24 months
  OS rate is defined as the proportion of patients who have not experienced death from any cause at 12 and 24 months after curative resection.
Adverse Events (AEs) | 24 months
  The grade of AEs and the number of patients with AEs are assessed based on CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No